CLINICAL TRIAL: NCT06202547
Title: Safety and Feasibility Study of Intra-ovarian Injection of Bone Marrow Mesenchymal Stromal Cells-derived Extracellular Vesicles in Idiopathic Premature Ovarian Failure Patients: Clinical Trial Phase I
Brief Title: Intra-ovarian Injection of MSC-EVs in Idiopathic Premature Ovarian Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 400000134; IRCT20080831001141N43 (Other: www.irct.ir)
Record Dates: First submitted 2023-12-05; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Premature Ovarian Failure
Keywords: Intra-ovarian injection; Mesenchymal stromal cells-derived extracellular vesicles
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intraovarian injection of MSC-EVs (Experimental): The patient is anesthetized and placed in a lithotomy position, after preparing and washing the vagina with normal saline, under transvaginal ultrasound guidance (Aloka-40000 vaginal probe, Japan) using needle puncture (Reproline medical Gmbh, Rheinbach/Germany). The injection of 2 ml of extracellular vesicles derived from MSCs (equivalent to 30 million cells) will be performed into one ovary of the patient (the accessible ovary).
  Interventions: Biological: Intra-ovarian injection of bone marrow mesenchymal stromal cells-derived extracellular vesicles

INTERVENTIONS:
Biological: Intra-ovarian injection of bone marrow mesenchymal stromal cells-derived extracellular vesicles — he patient is anesthetized and placed in a lithotomy position, after preparing and washing the vagina with normal saline, under transvaginal ultrasound guidance (Aloka-40000 vaginal probe, Japan) using needle puncture (Reproline medical Gmbh, Rheinbach/Germany). The injection of 2 ml of extracellular vesicles derived from MSCs (equivalent to 30 million cells) will be performed into one ovary of the patient (the accessible ovary).

SUMMARY:
Premature ovarian failure (POF) is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POF is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotrophins and low estradiol. The prevalence of POF is 1-2%. Extracellular vesicles (EVs) are membrane-packed vesicles that are secreted by a variety of cell types, including T cells, B cells, dendritic cells, platelets, mast cells, epithelial cells, endothelial cells, neuronal cells, cancerous cells, oligodendrocytes, Schwann cells, embryonic cells, and mesenchymal stromal cells-derived (MSCs). MSCs-EV more stable and induce stronger signaling and are produced in higher concentrations than stem cells. They demonstrate no inherent toxicity, are not associated with any long-term maldifferentiation of engrafted cells or tumor generation, and carry no apparent risk of aneuploidy or immune rejection following in vivo allogenic administration.Several studies have evaluated the safety and possible efficacy of injection MSCs-EV for the treatment of premature ovarian failure in animal models. Based on the available evidence, the study was designed with the aim of investigating the safety and effectiveness of intraovarian injection of MSCs-EV in patients with POF diagnosis.

DETAILED DESCRIPTION:
Investigating the effect of intraovarian injection of bone marrow-derived extracellular vesicles (MSC-EV) on serum levels of Follicle-Stimulating Hormone (FSH),Anti-Mullerian Hormone (AMH) levels, as well as the return of the menstrual cycle in infertile patients with premature ovarian failure, as well as the evaluation of its possible side effects. A before/after clinical trial (phase I) on 10 patients is designed. Eligible patients will be included in the study if they have written consent. Infertile women who have been diagnosed with premature ovarian failure and have normal body mass index and normal genetic tests are invited to participate in this project. Patients with early amenorrhea and certain immunological and cardiovascular diseases, as well as a history of ovarian masses or abnormal serological tests will not be included in the study. If the patient has undergone hormone replacement therapy (HRT), the HRT will be stopped for at least two months and then the injection cycle will be started.Injection of bone marrow-derived extracellular vesicles with a dose equivalent to 3 times 10 million clonal mesenchymal stem cells in 2 ml will be performed for all patients. Follow-up of patients in order to respond to treatment for 8 months based on evaluation of Follicle-Stimulating Hormone (FSH),Anti-Mullerian Hormone (AMH) levels, return of menstrual cycle, ovarian ultrasound and also check possible complications due to injection (fever, bacteremia, sepsis, Pelvic inflammatory disease, anaphylactic shock and hematoma from the first 24 hours and in the first week) will be done.

Primary Outcome Measures, Safety evaluation, [Time Frame: 8 months]:Early-onset possible side effects (fever, bacteremia, sepsis, PID, anaphylactic shock, and hematoma will be evaluated at the first 24 h and during the first week. Possible second side effects such as ovarian abscesses and benign or malignant neoplasms will be assessed until 8 months after intra-ovarian EV injection.

Secondary Outcome Measures, Feasibility evaluation, [Time Frame: 8 months]: The Serum FSH, Estradiol and AMH levels measurements and Return of menstrual cycle will be evaluated until months after intra-ovarian EV injection. Ultrasonography evaluation will be performed monthly to evaluate the ovarian volume (cc), the antral follicle count, Endometrium thickness, the number and size of the follicles.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20-38 years old
* Baseline serum level of follicle stimulating hormone (FSH) higher or equal to 25 IU/l at least twice with an interval of 3 or 4 months
* At least one year has passed since secondary amenorrhea and premature ovarian failure (POF) diagnosis
* Normal karyotype and fragile X messenger ribonucleoprotein 1 (FMR1) gene

Exclusion Criteria:

* Primary amenorrhea
* Congenital anomaly of the ovary
* Thyroid disease Immune system diseases such as lupus, etc.
* Previous and/or family history of ovarian tumor
* Previous and/or family history of suffering from major diseases in the past and present such as cancer
* Positive serological evidence regarding previous or current hepatitis B and C, Human T-lymphotropic virus 1, Human immunodeficiency virus (HIV), Syphilis Disturbance in the normal range of laboratory tests as levels of Hemoglobin Subunit Alpha 1 (HbA1), Alanine transaminase (ALT), The aspartate aminotransferase (AST), the number of white blood cells (WBCs), The creatinine (Cr), International normalised ratio (INR) , Platelets (Plt), Hematocrit (Hct) tests.
* History of specific systemic disease (rheumatology, endocrine, cardiovascular, etc.)
* Severe endometriosis (stage III and IV)
* Small and non-injectable ovaries Lack of patient satisfaction
* The patient's unwillingness to continue participating in the study

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Rate of ovary abscess | First 24 hours, first week and monthly up to 8 months after injection
  Sonographic evaluation of ovaries will be done for detection of ovarian abscess or any other ovarian lesion formation up to 8 months after intraovarian injection of extracellular vesicles derived from bone marrow mesenchymal stromal cells (any adverse events through follow-up visits (first 24 hours and first week after transplantation, 1, 2, 3, 4, 5, 6, 7 and 8 months after injection) will be checked and recorded.

SECONDARY OUTCOMES:
Basal follicle-stimulating hormone (FSH) serum level | Baseline,1 week as well as one, two, three, four , five, six, seven and eight months after transplantation
  Hormonal examination will be done with standard methods in the specialized laboratory of Royan Institute. A venous blood sample will be collected from all participants. The basal serum levels of FSH will be measured by Electrochemiluminescence immunoassay (ECLIA) using fully automated COBAS E-601 analyzer and a commercial kit (Roche Diagnostics GmbH, Mannheim, Germany). The Units of Measure will be presented as IU/l.
Serum anti-mullerian hormone (AMH) levels | Before the intervention (baseline) and also three, six and eight months after transplantation
  Hormonal examination will be done with standard methods in the specialized laboratory of Royan Institute. A venous blood sample will be collected from all participants. The basal serum levels of AMH will be measured by Electrochemiluminescence immunoassay (ECLIA) using fully automated COBAS E-601 analyzer and a commercial kit (Roche Diagnostics GmbH, Mannheim, Germany). The Units of Measure will be presented as ng/ml.
Menstruation recurrence rate | one, two, three, four , five, six, seven and eight months after transplantation
  Through monthly follow-up and asking the questions.The number of patients whose menstrual cycle has returned will be reported.
Antral follicle count | Before the intervention (baseline) as well as one, two, three, four , five, six, seven and eight months after transplantation
  Through monthly examination of specialized ultrasonography.The number of follicles measuring 2-10 mm in diameter observed in each ovary will be counted and recorded in the ultrasound examination.
The ovaries size and volume | One, two, three, four , five, six, seven and eight months after transplantation
  The Ovary size and volume will be determined through monthly examination of specialized ultrasonography. The volume estimate is calculated by the formula for an ellipsoid, where D1, D2, and D3 are the three axial measurements:
  D1 x D2 x D3 x 0.52

CONTACTS AND LOCATIONS:
Overall Officials: Faezeh Shekari, Ph.D, Principal Investigator — Department of Development of Stem Cell Sciences of Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran